CLINICAL TRIAL: NCT05642650
Title: Clinical Translational Research of Novel Wearable Device Based on Patented Sensing Technology in Non-Invasive Management of Heart Failure
Brief Title: Novel Wearable Device for Heart Failure Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingyi Ren, Professor of medicine(Cardiology), Deputy Director of the Cardiology Department and Director of the Heart Failure Center, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022-NHLHCRF-YXHZ-01
Record Dates: First submitted 2022-11-15; First posted 2022-12-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
Keywords: Novel Wearable Device; remote monitoring; Right heart catheterization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel wearable device strategy group (Experimental): Patients with a novel wearable device for monitoring and uploading data daily to collect monitoring data such as jugular vein pressure and exercise steps.
  Interventions: Device: novel wearable device
- Control group (No Intervention): Patients receive a standard of care for heart failure without a wearable device.

INTERVENTIONS:
Device: novel wearable device — Patients with a novel wearable device for monitoring and uploading data daily to collect monitoring data such as jugular vein pressure and exercise steps after discharge.
  Arms: Novel wearable device strategy group

SUMMARY:
Heart failure (HF) is a major cardiovascular disease with high readmission and mortality rate. A wearable device that could remotely monitor and detect the worsening HF early before the symptoms appear will help reduce HF readmissions effectively. The purpose of the current study is to examine the efficiency of a novel wearable device based on flexible strain sensor comparing to the clinical 'gold standard,' and then transform it into a clinical application.

DETAILED DESCRIPTION:
The prospective cohort study aims to examine the efficiency of a novel wearable device based on a flexible strain sensor to improve the outcomes of patients with HF compared to the standard-of-care without wearable device monitoring.

The primary and secondary endpoints will be examined in subgroups determined by baseline variables reflecting demography,NYHA functional class,left ventricular ejection fraction,natriuretic peptide,additional co-morbidities,and others.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HF ≥ 3 months
2. Diagnosis of NYHA Class III HF
3. Subjects with age ≥ 18 years
4. At least 1 HF hospitalization within 12 months prior to enrollment
5. Subjects with elevated ambulatory levels of BNP/NT-proBNP

Exclusion Criteria:

1. Subjects unable to cooperate to complete the trial.
2. Subjects with severe arrhythmia.
3. Subjects with cardiac shock.
4. Subjects with acute myocardial infarction.
5. Subjects with local skin infections and injuries in the jugular vein area
6. Subjects with active uncontrolled infections
7. Subjects with eGFR < 25 mL/min/1.73m2
8. Pregnant women, or women likely to undergo pregnancy
9. Subjects with life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-02-07 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Hospital Readmissions for Heart Failure | Up to 6 months
  Total hospitalizations for heart failure will be monitored via follow-up.

SECONDARY OUTCOMES:
Concordance of the Jugular Vein Pressure with the RHC Measurement | Up to 6 months
  Accuracy of jugular vein pressure measurements by the novel wearable device compared to right heart catheterization.
Change From Baseline N-terminal Pro-brain Natriuretic Peptide(NT-proBNP) or Brain Natriuretic Peptide(BNP) | Up to 6 months
  Change from baseline to 6 months in N-terminal pro-brain natriuretic peptide (NT-proBNP) or Brain Natriuretic Peptide(BNP). NT-proBNP/BNP level will be measured using commercial kits system during the follow-up period. Change from baseline was defined as the value of NT-proBNP/BNP at 6 months minus the baseline value. Baseline value was defined as the mean of all available measurements from the screening visit.
Change in Exercise Capacity as Measured by the 6-Minutes-Walking-Test (6MWT) Distance. | Up to 6 months
  Change from baseline to 6 months in exercise capacity as measured by the distance walked in 6 minutes in standardised conditions.
Compliance Percentage of Patients | Up to 6 months
  Patient adherence to daily measurement and transmission of sensor readings will be recorded.
Change in Quality of Life | Up to 6 months
  Quality of life will be measured with the Kansas City Cardiomyopathy Questionnaire (KCCQ) answered by the patients directly on a patient application.KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The KCCQ total symptom score incorporates the symptom domains into a single score. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Change in New York Heart Association (NYHA) functional class. | Up to 6 months
  NYHA class will be evaluated according to the patients' clinical characteristics during the follow-up.NYHA Functional Classification places patients in one of four categories based on how much they are limited during physical activity; Class I being best and Class IV being the worst functional class. Class I has no limitation to physical activity, Class II has slight limitation to physical activity, Class III has marked limitation of physical activity, and Class IV is unable to carry out any physical activity without severe discomfort.
Freedom From a Device/System-related Complication | Up to 6 months
  Device/System-related Complications refer to adverse events such as device failure and allergy.

OTHER OUTCOMES:
Subjects Included the Endpoint of Cardiovascular Mortality | Up to 6 months
  Rate of cardiovascular mortality will be monitored via follow-up.
Subjects Included the Endpoint of all-cause Mortality | Up to 6 months
  Rate of all-cause mortality will be monitored via follow-up.

IPD SHARING:
Plan to Share IPD: No